CLINICAL TRIAL: NCT00213928
Title: A Single-blind, Randomized Trial of Horse Chestnut Seed Extract for the Treatment of Lymphedema of the Arm in Breast Cancer Survivors
Brief Title: Horse Chestnut Seed Extract for Lymphedema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2004-050; CC 01106 (Other: IRB# 2002-050)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2011-07

CONDITIONS: Lymphedema of Arm
MeSH Terms: interventions — horse chestnut seed

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Horse Chestnut Seed Extract (Active Comparator): Horse chestnut seed extract (escins, aesins)
  Interventions: Drug: Horse Chestnut Seed Extract

INTERVENTIONS:
Drug: Horse Chestnut Seed Extract — Control (no intervention) vs Horse Chestnut Seed Extract
  Arms: Horse Chestnut Seed Extract

SUMMARY:
To help Treat Lymphedema of the Arm in Breast Cancer Survivors with Horse chestnut Seed Extract

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the effectiveness of escin (as horse chestnut seed extract) for arm lymphedema in women following treatment for breast cancer, to evaluate the accuracy and sensitivity of bioelectric impedance as a measurement of lymphedema of the arm, and to validate the proposed arm lymphedema quality-of-life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patient demonstrates unilateral (ipsilateral to breast cancer resection side) lymphedema of the upper extremity. An extravascular water ratio of ³1.1/1 between the affected vs normal arm using multiple-frequency bioelectric impedance will be used as a criterion for lymphedema. There is not upper limit to the extent of arm volume (lymphedema)
* Patient is greater than 6 months from last surgical and/or radiation treatment to the affected axilla.

Exclusion Criteria:

* Patients may not be receiving or be scheduled to receive cytotoxic or radiation chemotherapy treatment while on this lymphedema study (Last chemotherapy > 4 weeks prior). Women who are being treated adjuvantly with tamoxifen, raloxifene, or an aromatase inhibitor remain eligible
* Patients with a history of recurrent (more than 1 episode) arm cellulitis, prior or existing venous clot, or considered to have "woody" fibrosis of the affected arm are not eligible. Antibiotics used to treat any prior episode of cellulitis must have be completed no more recently than 3 months prior to initial screening.

Min Age: 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2002-05; Primary Completion 2004-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Reduction of arm lymphedema

SECONDARY OUTCOMES:
- comparison of bioelectric impedance to measure lymphedema changes
- validation of bioelectric impedance to measure lymphedema changes
- validation of lymphedema questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Hutson, PharmD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States